CLINICAL TRIAL: NCT06514976
Title: Multi-center International Observational Study of Efficiency of the Drug Cytoflavin®, Solution for Infusions in Patients With Ischemic Stroke Not Receiving Reperfusion Therapy.
Brief Title: Observational Study of Efficiency of Cytoflavin, in Patients With Ischemic Stroke Not Receiving Reperfusion Therapy
Status: Recruiting | Type: Observational
Sponsor: POLYSAN Scientific & Technological Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Other Study IDs: CTF-NIS-2024
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2024-07

CONDITIONS: Stroke, Acute; Stroke, Ischemic
Keywords: stroke; сytoflavin
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — cytoflavin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- The test group: Basic therapy + Cytoflavin
  Interventions: Drug: Cytoflavin
- The control group: Basic therapy (with or without other neuroprotector)

INTERVENTIONS:
Drug: Cytoflavin — Cytoflavin solution for infusions. 20-40 ml/day (10 ml with the interval of 8-12 hours for 10 days; the single dose is increased up to 20 ml in case of the severe form of the disease) by intravenous drop infusion in dilution per 100-200 ml of 0.9% sodium chloride solution for 10 days; rate of administration: 3-4 ml/min
  Groups: The test group

SUMMARY:
Stroke remains one of the main socially significant problems in the healthcare in the third millennium. The lethality in persons with history of stroke by the end of the 1st year of disease is high. A trend to increased frequency of stroke in the young age is observed during the last decade; third of patients is working-age individuals, out of whom only 15-20% returns to labor, and others remain disabled persons requiring constant medical and social support

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form
2. Age from 18 years and older
3. Diagnosis: Acute cerebrovascular accident of ischemic type (ischemic stroke) developed within 36 hours before enrollment in the study
4. Motor neurologic deficit measurable using the NIHSS Scale (score for item 5 and/or 6 at the time of starting the therapy ≥ 1))
5. Conservative stroke treatment tactics (without reperfusion therapy thrombolysis/thrombus extraction)
6. According to the routine clinical practice, the patient is scheduled to receive the treatment as per one of the following regimens:

   * Cytoflavin® 20-40 ml/day as a course of not less than 10 days or
   * another neuroprotector - course of not less than 10 days (or without neuroprotector)

Exclusion Criteria:

1. NIHSS 1a (coma) score 3 at the time of enrollment
2. Initial severe disablement (corresponding to mRS > 2) requiring external assistance in everyday life before development of stroke
3. History of Parkinson's disease, dementia, multiple sclerosis, and other significant diseases accompanied by neurologic deficit
4. Severe comorbidity with expected lifespan of not more than 6 months
5. Pregnancy and breastfeeding
6. Any other concomitant medical or serious psychic conditions, which make the patient ineligible for participation in the study, restrict lawfulness of obtaining the informed consent, or can influence the patient's ability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged above 18 years with diagnosis of ACVA of ischemic type who did not receive and are not scheduled for reperfusion therapy (thrombolysis, thrombus extraction).
Sampling Method: Probability Sample
Enrollment: 562 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with favorable functional outcome (score 0-2) according to Modified Rankin Scale (mRS) on Day of Discharge (assessment at Visit 4 or Visit 5, on Day of Discharge) and on Day 90; | Base, day 14, day 21, day 90
  Modified Rankin Scale (mRS)

SECONDARY OUTCOMES:
Total score according to Modified Rankin Scale (mRS) on Day of Discharge and Day 90 in the test and control group; | Day 14, day 21, day 90
  Modified Rankin Scale (mRS)
Total score according to Rivermead Scale on Day 7, Day 14, Day 21, and Day 90 in the test and control group | Day 7, day 14, day 21, day 90
  Rivermead Scale
Change of the total score according to National Institute of Health Stroke Scale (NIHSS) on Day 3, Day 7, Day 14, and Day 21 as compared to the baseline level (Day 1); | Day 7, day 14, day 21, day 90
  National Institute of Health Stroke Scale (NIHSS)
Change of the total score according to Stroke-Specific Quality of Life Scale (SS-QOL) on Day 90 as compared to Day of Discharge; | Day 14, day 21, day 90
  Stroke-Specific Quality of Life Scale (SS-QOL)
Percentage of patients with repeated ACVA or TIA during the study; | Day 90
  Repeated ACVA or TIA
Percentage of patients with lethal outcome in the period of hospitalization and follow-up | Day 90
  Lethal outcome

CONTACTS AND LOCATIONS:
Locations (17):
- Russia (17):
  - "Ivanovo Regional Clinical Hospital", Ivanovo
  - Kazan State Medical University, Kazan'
  - State Autonomous Institution of Health Interregional clinical diagnostic center, Kazan'
  - Moscow City Clinical Hospital No.64 (CCH named after V.V. Vinogradov), Moscow
  - N.I. Pirogov City Clinical Hospital No. 1, Moscow
  - Vorohobov's City Clinical Hospital №67, Moscow
  - City Clinical Hospital No. 1 Novosibirsk, Novosibirsk
  - Alexandrovskaya hospital, Saint Petersburg
  - Almazov National Medical Research Centr, Saint Petersburg
  - City Mariinsky Hospital, Saint Petersburg
  - Nikolaevskaya Hospital, Saint Petersburg
  - Saint-Petersburg I. I. Dzhanelidze research institute of emergency medicine, Saint Petersburg
  - St. Petersburg State Budgetary Institution of Public Health "City Hospital No. 40 of Kurortny District", Saint Petersburg
  - The City Hospital of the Holy Martyr Elizabeth, Saint Petersburg
  - Smolensk Regional Clinical Hospital, Smolensk
  - Municipal Clinical Hospital #13, the City of Ufa, State Budgetary Healthcare Institution of the Republic of Bashkortostan, Ufa
  - Budgetary healthcare institution of the Voronezh region "Voronezh Regional Clinical Hospital No. 1", Voronezh